CLINICAL TRIAL: NCT04387799
Title: Major Determinants of COVID-19 Associated Pneumonia
Brief Title: Determinants of COVID-19 Pneumonia (MC-19)
Acronym: MC-19
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Associate Professor of Internal Medicine, Catholic University of the Sacred Heart
Other Study IDs: 20200505
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Pneumonia, Viral; Pneumonia, Bacterial; Coronavirus Infection; Obstructive Lung Disease
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia, Bacterial; Coronavirus Infections; Lung Diseases, Obstructive | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative PCR Covid associated Pneumonia: Patients with pneumonia who test negative to RT-PCR
  Interventions: Diagnostic Test: Serology for Covid-19
- Positive PCR Covid associated Pneumonia: Patients with pneumonia from Covid 19

INTERVENTIONS:
Diagnostic Test: Serology for Covid-19 — Antibody tests designed to provide results to individuals or healthcare providers can show whether someone was previously infected with SARS-CoV-2 being the RT-PCR negative for the population of patients
  Groups: Negative PCR Covid associated Pneumonia

SUMMARY:
Molecular testing (e.g PCR) of respiratory tract samples is the recommended method for the identification and laboratory confirmation of COVID-19 cases.

Recent evidence reported that the diagnostic accuracy of many of the available RT-PCR tests for detecting SARS-CoV2 may be lower than optimal.

Of course, the economical and clinical implications of diagnostic errors are of foremost significance and in case of infectious outbreaks, namely pandemics, the repercussions are amplified. False positives and false-negative results may jeopardize the health of a single patient and may affect the efficacy of containment of the outbreak and of public health policies.

In particular, false-negative results contribute to the ongoing of the infection causing further spread of the virus within the community, masking also other potentially infected people.

DETAILED DESCRIPTION:
As demonstrated by a study conducted by Ai et al., including 1014 suspect COVID-19 cases who underwent multiple RT-PCR testing and chest-CT, overall 88% of patients had positive CT scans while RT-PCR positivity was found only in 59% of all cases. Also, as reported by Yang et al, the total positive rate of RT-PCR for throat swab samples was reported to be about 30% to 60% at initial presentation. Thus, a negative result does not exclude the possibility of infection and should not be used as the only criterion for treatment of patient and management decisions.

Reasons for false negative RT-PCR may include the lack of identification or inadequate procedures for specimen collection, handling and storage, as well as active viral recombination or testing carried out of the diagnostic window.

From preliminary studies has emerged that patients may show very early but significant CT changes even before RT-PCR studies. Hence, the necessity for developing a combined approach for the diagnosis of these particular patients who present with negative RT-PCR test results.

The investigators hypotheses is that several patients who presented with pneumonia confirmed at CT scan during the Coronavirus outbreak, and who tested negative for SARS-CoV2 at RT-PCR could probably be affected by the disease and need to be carefully observed.

Primary end-point The primary end-point of our prospective, observational study is to assess if inpatients who presented with pneumonia but had a negative test for Covid-19 are positive at the serology for SARS-CoV-2.

Secondary end-points Among the other secondary end-points, the investigators aim is to find if the combination of CT scan and serology could help in the identification of those patients who were initially negative at laboratory testing alone.

Other secondary end-points are the efficacy of different pharmaceutical treatments against Covid-19 that were empirically started in those highly suspicious cases and the development of an approach useful for those patients who initially tested negative for Covid-19 infection.

Methods Before starting the study, the protocol will be submitted to and approved by the local Ethical Committees at the Fondazione Policlinico Universitario A. Gemelli IRCCS, Catholic University, Rome, Italy. Before enrollment each subject will sign the informed consent.

Inclusion criteria: hospitalized subjects of both sexes aged 18 years or older with diagnosis of pneumonia, confirmed by chest imaging and oxygen saturation (SaO2) ≤ 94% in ambient air, Covid-19 test negative, given informed consent to data collection from the patient or from the patient's legal representative if the patient is too unwell to provide consent.

Exclusion criteria: age lower than 18 years, pregnancy or breast-feeding. Nasopharyngeal swab samples will be taken for quantitative real-time polymerase chain reaction to make diagnosis of Covid19 (2 repeated tests).

Data collected include time of symptoms (cough, fever, dyspnea, conjunctivitis, diarrhea, asthenia, arthralgia) age, sex, height, weight, education, alcohol and smoking habits, morbidities, plasma glucose, creatinine, transaminases, γ-GT, total cholesterol, HDL-cholesterol, triglycerides, complete blood count, D-dimer, lactic acid dehydrogenase (LDH), high-sensitivity C-reactive protein (hs-CRP), creatinkinase (CK), ferritin, HbA1c, chest X rays, chest CT scan, cultures, therapy for pneumonia, other treatments including anti-hypertensive and anti-hyperglycemic agents, body temperature, blood pressure, and oxygen flow rate or other types of oxygen treatment.

Five ml of plasma divided in aliquots of 1 ml each will be also obtained and stored at -80°C in anonymized way for future analysis, including third parties.

Sample size If there is truly no difference between the standard and experimental treatment (16% in both groups), then 260 patients are required to be 90% sure that the limits of a two-sided 90% confidence interval will exclude a difference between the standard and experimental group of more than 15% Significance (α) = 0.05 Power (1-β)= 90% Percentage deaths in both control and experimental group = 16% Equivalence limit = 15%

Calculation based on the formula:

n = 2 × f(α, β/2) × π × (100 - π) / d2 where π is the true percent 'success' in both the control and experimental treatment groups, and f(α, β) = [Φ-1(α) + Φ-1(β)]2 Φ-1 is the cumulative distribution function of a standardised normal deviate.

Statistics The association between recovery and patient groups will be tested by means of a Fisher exact test. A Cox Proportional-Hazard regression will be used to compare survival curves (times to improvement) among the studied groups by correcting for the administered therapy and for all the quantitative collected variables. Quantitative variables, measured at hospital admission, will be compared among groups using ANOVA. In univariable analyses, categorical variables, as gender, education, alcohol consumption and smoke habits will be analysed by means of a Chi-Squared test to study their association with the recovery, while a logistic regression model will be used to test possible quantitative predictors of recovery. A multivariable logistic model, with a stepwise selection procedure, will be then used to test all the variables that are significant in a univariable analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pneumonia; Covid-19 test negative; hospitalized subjects; both sexes; given informed consent

Exclusion Criteria:

* age lower than 18 years; pregnancy; breast-feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects hospitalized for pneumonia who tested negative at RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Serology | 3 weeks
  assess if inpatients who presented with pneumonia but had a negative test for Covid-19 are positive at the serology for SARS-CoV-2.

SECONDARY OUTCOMES:
Efficacy of CT scan and Serology | 3 weeks
  to find if the combination of CT scan and serology could help us in the identification of those patients who were initially negative at laboratory testing alone.
Efficacy of different pharmaceutical treatments | 3 weeks
  the efficacy of different pharmaceutical treatments against Covid-19

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Background] Lippi G, Simundic AM, Plebani M. Potential preanalytical and analytical vulnerabilities in the laboratory diagnosis of coronavirus disease 2019 (COVID-19). Clin Chem Lab Med. 2020 Jun 25;58(7):1070-1076. doi: 10.1515/cclm-2020-0285. PMID 32172228
- [Background] Lippi G, Plebani M, Graber ML. Building a bridge to safe diagnosis in health care. The role of the clinical laboratory. Clin Chem Lab Med. 2016 Jan;54(1):1-3. doi: 10.1515/cclm-2015-1135. No abstract available. PMID 26630697
- [Background] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Background] Xie X, Zhong Z, Zhao W, Zheng C, Wang F, Liu J. Chest CT for Typical Coronavirus Disease 2019 (COVID-19) Pneumonia: Relationship to Negative RT-PCR Testing. Radiology. 2020 Aug;296(2):E41-E45. doi: 10.1148/radiol.2020200343. Epub 2020 Feb 12. PMID 32049601
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261